CLINICAL TRIAL: NCT05727306
Title: Healthcare Disparities in Alopecia Areata: UK Population-based Cohort Study
Brief Title: Healthcare Disparities in Alopecia Areata
Status: Completed | Type: Observational
Sponsor: Momentum Data (Industry)
Collaborators: Pfizer (Industry); University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: p068
Record Dates: First submitted 2023-01-11; First posted 2023-02-14 (Actual); Results first posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-05

CONDITIONS: Alopecia Areata
MeSH Terms: conditions — Alopecia Areata

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- People with Alopecia Areata: Children and adults aged 12+ with new onset Alopecia Areata registered with a contributing General practitioner (GP) practice during the study period.
  Interventions: Other: No intervention
- People without Alopecia Areata: Children and adults aged 12+ without Alopecia Areata registered with a contributing GP practice during the study period.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Observational analysis of usual care only.

SUMMARY:
Alopecia areata (AA) is a common immune-mediated non-scarring alopecia often associated with substantial morbidity. There are however, limited population-based data on potential disparities in the burden of AA, including across people of different ethnicities and deprivation.

We aimed to provide the first large-scale, population-based estimate of lifetime risk of AA overall and by important sociodemographic subgroups. As AA is associated with an increased burden of mental health conditions and work-related outcomes (unemployment, time off work), a detailed understanding of the burden of disease in different sociodemographic groups is vital to plan resource provision.

DETAILED DESCRIPTION:
The overall purpose of the study is to provide an estimate of the cumulative lifetime incidence of AA in the population overall and by important sociodemographic groups. Moreover, to do a subgroup analysis in the AA population to identify health-related disparities across people in different socioeconomic strata, geographical distribution, sex and ethnic groups. The disparities that will be considered are AA associated: Mental health conditions; healthcare utilisation; and work impact (time off work and unemployment).

The cumulative lifetime risk of AA was estimated at age 80 years (approximate life expectancy in the UK) using survival models, with age as the timescale and accounting for the competing risk of death.

The assessment of any associations with baseline characteristics and the outcomes of interest will be assessed using Cox proportional hazards models (time to event outcomes) and Poisson regression (repeated event outcomes) models.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged greater than 12 over the study period.
* Registered with the contributing primary care practice for any duration during the study period

Exclusion Criteria:

* People diagnosed with AA before the study period.

Ages: 12 Years to 95 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All individuals with new onset AA during the study period defined by the presence of at least one disease specific diagnostic code will be eligible for inlcusion in the AA cohort. Controls will be matched people without AA matched on age, sex, geography, ethnicity, socioeconomic status.
Sampling Method: Non-Probability Sample
Enrollment: 4052231 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-07-24 (Actual); Study Completion 2024-08-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew McGovern, MD, Study Director — Momentum Data
Locations (1):
- Momentum Data Limited, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Individual patient data is confidential but can be made available in an anonymised form to bone fide researchers subject to the required data protection training and other requirements. All data will remain behind a firewall and will only be available for access through a secured computer network.
Supporting Information: SAP
Time Frame: There is no pre-specified time-frame for data availability; this will be considered on an individual basis for each request.
Access Criteria: As above.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 4,052,231 adults and children (aged 12+) in the final study population, 6,183 people who developed Alopecia Areata (AA) between 1 January 2009 and 31 December 2018 were matched to 24,718 people without AA.
Pre-assignment Details: People that did not develop Alopecia Areata but had a diagnosis of a nonspecific or alopecia alternative condition, or less than 12 months of follow-up available, were excluded from the study.
Period: Overall Study
Arm/Group | People With Alopecia Areata | People Without Alopecia Areata
Started | 6183 | 24718
Aged 18-65 Years Old | 5293 | 20864
Completed | 6183 | 24718
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | People With Alopecia Areata | People Without Alopecia Areata | Total
Number analyzed (Participants) | 6183 | 24718 | 30901
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 35 [26 to 47] | 35 [25 to 47] | 35 [25 to 47]
Age, Customized [Count of Participants; unit: Participants]
  12-17 | 529 | 2111 | 2640
  18-29 | 1699 | 6792 | 8491
  30-49 | 2666 | 10659 | 13325
  50+ | 1289 | 5156 | 6445
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3342 | 13366 | 16708
  Male | 2841 | 11352 | 14193
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 3205 | 12820 | 16025
  Black | 241 | 960 | 1201
  Asian | 1129 | 4515 | 5644
  Other | 264 | 1047 | 1311
  Not recorded | 1344 | 5376 | 6720
Geographic area: Urban, Rural [Count of Participants; unit: Participants]
  Urban | 5150 | 20590 | 25740
  Rural | 913 | 3648 | 4561
  Not recorded | 120 | 480 | 600
Index of multiple deprivation (IMD) [Count of Participants; unit: Participants] — Index of Multiple Deprivation (IMD) is a United Kingdom (UK) national deprivation measure of deprivation which is based on the patient postcode. IMD has been stratified into quintiles with IMD 1 representing most deprived and IMD 5 being the least deprived.
  Participants
    1 (most deprived) | 1339 | 5356 | 6695
    2 | 1277 | 5108 | 6385
    3 | 1091 | 4356 | 5447
    4 | 1144 | 4573 | 5717
    5 (least deprived) | 1205 | 4818 | 6023
    Not recorded | 127 | 507 | 634
Body Mass Index (BMI), Categorical [Count of Participants; unit: Participants]
  < 18.5 Underweight | 315 | 1303 | 1618
  18.5-25 Normal weight | 2277 | 8842 | 11119
  25-30 Overweight | 1644 | 5901 | 7545
  30-35 Class I obesity | 665 | 2664 | 3329
  35-40 Class II obesity | 245 | 941 | 1186
  40+ Class III obesity | 132 | 496 | 628
  Not recorded | 905 | 4571 | 5476
Smoking status [Count of Participants; unit: Participants]
  Non-smoker | 2538 | 11676 | 14214
  Active smoker | 1868 | 5561 | 7429
  Ex-smoker | 1529 | 5741 | 7270
  Not recorded | 248 | 1740 | 1988
Alcohol status [Count of Participants; unit: Participants]
  Non-drinker | 1272 | 4628 | 5900
  Safe use | 2750 | 10927 | 13677
  Hazardous use | 686 | 2596 | 3282
  Alcoholism | 117 | 314 | 431
  Not recorded | 1358 | 6253 | 7611
Geographical region [Count of Participants; unit: Participants]
  London | 1488 | 5952 | 7440
  East Midlands | 227 | 904 | 1131
  East of England | 253 | 1009 | 1262
  North East | 209 | 833 | 1042
  North West | 1160 | 4640 | 5800
  South East | 1053 | 4212 | 5265
  South West | 635 | 2540 | 3175
  West Midlands | 417 | 1665 | 2082
  Yorkshire and The Humber | 614 | 2456 | 3070
  Not recorded | 127 | 507 | 634

OUTCOME MEASURES:

1. Primary Outcome: Likelihood of Depressive Episodes
Description: Estimated using logistic regression and reported using adjusted odds ratios
Time Frame: Data was collected retrospectively, assessed prior to and up to two years following initial Alopecia Areata diagnosis for each participant
Measure: Count of Participants; unit: Participants
Groups:
- People Without Alopecia Areata (Reference Group): Children and adults aged 12+ without Alopecia Areata registered with a contributing GP practice during the study period.
  No intervention: Observational analysis of usual care only.
Arm/Group | People With Alopecia Areata | People Without Alopecia Areata (Reference Group)
Number analyzed (Participants) | 6183 | 24718
Participants | 1217 | 3576
Statistical Analysis 1: Comparison: People Without Alopecia Areata (Reference Group); Test type: Superiority; Odds Ratio (OR) = 1.35, 95% CI 2-sided [1.25 to 1.46] — Calculated as the odds of having a depressive episode in participants diagnosed of Alopecia Areata vs. participants without Alopecia Areata. Odds Ratio adjusted for sociodemographic, clinical characteristics and major comorbidities

2. Primary Outcome: Likelihood of Recurrent Major Depressive Disorder
Description: Estimated using logistic regression and reported using adjusted odds ratios
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- People Without Alopecia Areata (Reference Gropup): Children and adults aged 12+ without Alopecia Areata registered with a contributing GP practice during the study period.
  No intervention: Observational analysis of usual care only.
Arm/Group | People With Alopecia Areata | People Without Alopecia Areata (Reference Gropup)
Number analyzed (Participants) | 6183 | 24718
Participants | 835 | 2264
Statistical Analysis 1: Comparison: People Without Alopecia Areata (Reference Gropup); Test type: Superiority; Odds Ratio (OR) = 1.45, 95% CI 2-sided [1.32 to 1.58] — Calculated as the odds of having recurrent depressive disorder in participants diagnosed of Alopecia Areata vs. participants without Alopecia Areata. Odds Ratio adjusted for sociodemographic, clinical characteristics and major comorbidities

3. Primary Outcome: Likelihood of Anxiety Disorder
Description: Estimated using logistic regression and reported using adjusted odds ratios
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | People With Alopecia Areata | People Without Alopecia Areata (Reference Group)
Number analyzed (Participants) | 6183 | 24718
Participants | 1113 | 3188
Statistical Analysis 1: Comparison: People Without Alopecia Areata (Reference Group); Test type: Superiority; Odds Ratio (OR) = 1.40, 95% CI 2-sided [1.30 to 1.51] — Calculated as the odds of having anxiety in participants diagnosed of Alopecia Areata vs. participants without Alopecia Areata. Odds Ratio adjusted for sociodemographic, clinical characteristics and major comorbidities

4. Secondary Outcome: Relative Incidence of Primary Care Attendances
Description: Estimated using negative binomial regression and reported as adjusted incidence rate ratio
Time Frame: Data was collected retrospectively, assessed up to two years following initial Alopecia Areata diagnosis for each participant
Measure: Number; unit: Count of primary care visits
Groups:
- People Without Alopecia Areata (Reference Group): Children and adults aged 12+ without Alopecia Areata registered with a contributing GP practice during the study period (reference group).
  No intervention: Observational analysis of usual care only.
Arm/Group | People With Alopecia Areata | People Without Alopecia Areata (Reference Group)
Number analyzed (Participants) | 6183 | 24718
Count of primary care visits | 39034 | 109052
Statistical Analysis 1: Comparison: People Without Alopecia Areata (Reference Group); Test type: Other; Incidence rate ratio (IRR) = 1.42, 95% CI 2-sided [1.37 to 1.46] — Calculated as the incidence rate of attending primary care in participants diagnosed of Alopecia Areata vs. participants without Alopecia Areata. Incidence rate ratio adjusted for sociodemographic, clinical characteristics and major comorbidities

5. Secondary Outcome: Relative Incidence of Dermatology Referrals
Description: Estimated using Cox proportional hazard regression and reported as Adjusted hazard ratio
Time Frame: as for outcome 4
Measure: Number; unit: Count of dermatology referrals
Arm/Group | People With Alopecia Areata | People Without Alopecia Areata (Reference Group)
Number analyzed (Participants) | 6183 | 24718
Count of dermatology referrals | 1352 | 743
Statistical Analysis 1: Comparison: People Without Alopecia Areata (Reference Group); Test type: Other; Hazard Ratio (HR) = 8.26, 95% CI 2-sided [7.55 to 9.04] — Calculated using Cox Proportional Hazard model.Reflects a comparison of incidence rates between participants diagnosed with Alopecia Areata (AA) and those without AA. Adjusted for sociodemographic,clinical characteristics and major comorbidities

6. Secondary Outcome: Relative Incidence Psychological Therapy
Description: Estimated using Cox proportional hazard regression and reported as adjusted hazard ratio
Time Frame: as for outcome 4
Measure: Number; unit: Count of therapy visits
Arm/Group | People With Alopecia Areata | People Without Alopecia Areata (Reference Group)
Number analyzed (Participants) | 6183 | 24718
Count of therapy visits | 248 | 672
Statistical Analysis 1: Comparison: People Without Alopecia Areata (Reference Group); Test type: Other; Hazard Ratio (HR) = 1.36, 95% CI 2-sided [1.17 to 1.57] — [estimate comment as in outcome 5, analysis 1]

7. Secondary Outcome: Relative Incidence of Unemployment
Description: Unemployment identified by issue of IB113 or ESA113 forms for unemployment. Relative incidence estimated using Cox proportional hazard regression and reported as Adjusted hazard ratio
Time Frame: as for outcome 4
Measure: Number; unit: Count of unemployment forms issued
Groups:
- People With Alopecia Areata: Adults aged 18-65 with new onset Alopecia Areata registered with a contributing General practitioner (GP) practice during the study period.
  No intervention: Observational analysis of usual care only.
- People Without Alopecia Areata (Reference Group): Adults aged 18-65 without Alopecia Areata registered with a contributing GP practice during the study period (reference group).
  No intervention: Observational analysis of usual care only.
Arm/Group | People With Alopecia Areata | People Without Alopecia Areata (Reference Group)
Number analyzed (Participants) | 5293 | 20864
Count of unemployment forms issued | 89 | 209
Statistical Analysis 1: Comparison: People Without Alopecia Areata (Reference Group); Test type: Other; Hazard Ratio (HR) = 1.46, 95% CI 2-sided [1.14 to 1.87] — [estimate comment as in outcome 5, analysis 1]

8. Secondary Outcome: Relative Incidence of Time Off Work
Description: Time off work identified by recorded issue of Med 3 certificate in primary care. Relative incidence estimated using Cox proportional hazard regression and reported as Adjusted hazard ratio
Time Frame: as for outcome 4
Measure: Number; unit: Count of Med 3 certificates issued
Arm/Group | People With Alopecia Areata | People Without Alopecia Areata (Reference Group)
Number analyzed (Participants) | 5293 | 20864
Count of Med 3 certificates issued | 884 | 2268
Statistical Analysis 1: Comparison: People Without Alopecia Areata (Reference Group); Test type: Other; Hazard Ratio (HR) = 1.49, 95% CI 2-sided [1.38 to 1.61] — [estimate comment as in outcome 5, analysis 1]

ADVERSE EVENTS:
Description: Deaths, serious adverse events, and nonserious adverse events were not assessed for study participants.
Arm/Group | People With Alopecia Areata | People Without Alopecia Areata
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan: Study Protocol (2022-11-02): https://cdn.clinicaltrials.gov/large-docs/06/NCT05727306/Prot_SAP_001.pdf